CLINICAL TRIAL: NCT06589960
Title: Effect of Lifestyle Modification on Patients with Knee Osteoarthritis Attending NRC Rheumatology Clinic
Brief Title: Effect of Lifestyle Modification on Patients with Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 8/4/7
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2022-10

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Lifestyle; Modification; WOMAC
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): * Health education
  * Physical exercise
  Interventions: Combination Product: Health education and physical exercise

INTERVENTIONS:
Combination Product: Health education and physical exercise — Nine face to face sessions and group discussion health education sessions. An Educational booklet was prepared and distributed to all attendants.
  Lab results were discussed individually with each participant.
  Rheumatologist and physiotherapist also provided messages.
  The exercise program targeted and strengthened the muscles around the knee especially quadriceps muscle, stretching the muscles of lower limbs, and stretching and increasing the range of motion of front and back lower limb muscles (quadriceps muscle, hamstring muscle, gluteus muscle and calf muscles).
  Phone calls to follow up the participants and maximize their adherence to the health education program. WhatsApp groups was created, and messages were distributed to summarize the content of the booklet and the exercises videos.
  Final reassessment to assess the effect of health education and lifestyle modification was carried out with participants who continued till the end of the study.

SUMMARY:
This is a cross-sectional study carried out on 180 Knee osteoarthritis (KOA) patients who were consecutively recruited from the Rheumatology Outpatient Clinic at National Research Center (NRC), Egypt. A face-to-face interview was carried out to collect data about demographic data, medical history, and Knowledge, Attitude and Practice (KAP). Assessment of symptoms, disease severity, and physical disability was carried out using Western Ontario and McMaster Universities Arthritis Index (WOMAC). Quality of life was also assessed using Osteoarthritis Knee and Hip Quality of Life (OAKHQOL) questionnaire. The studied participants were subjected to clinical examination and anthropometric measurements and a blood sample was collected from them to measure inflammatory biomarkers Interleukin-6 (IL-6). Then a health education and physical exercise were done. An Educational Booklet was designed and distributed to the studied patients. WOMAC, OAKHQOL, and KAP questionnaires were used to assess the effect of health education and lifestyle modification on the participants.

DETAILED DESCRIPTION:
I) Pre-intervention was done by:

1. Sociodemographic questionnaire: to gather information regarding participants age, gender, marital status, occupation, level of education, smoking habits, duration of the disease, medical history and medications taken.
2. Osteoarthritis Knee and Hip Quality of Life (OAKHQOL) questionnaire: The OAKHQOL is a specific tool to measure QOL in knee and hip OA as it takes into account specific themes that are exclusive to the QOL of patients with knee and hip OA (social support, sleep, side effects of drugs, plans for the future, embarrassment to be seen by people, use of public transport, difficulty in moving after staying in the same position, and sexuality). The concept of this questionnaire was based on the World Health Organization definition of QOL. It is a self-administered questionnaire the original questionnaire was developed in French and later in English, while in the current study, it was translated by the researcher into the Arabic language. It has 43 items which fall into five domains: physical activity (16 items), mental health (13 items), pain (4 items), social support (4 items), social functioning (3 items), and three items are independent. Response to all items is by a Numerical Rating Scale (NRS) (0-10). A total score for each subscale is calculated by averaging the values for items of the same dimension and is normalized to a score from 0 (worst HRQOL) to 100 (best HRQOL). Evaluation of the OAKHQOL has shown the reliability of the five domains to be satisfactory (interclass correlation coefficients: 0.70-0.85), the construct validity to be adequate (Spearman correlation coefficients: 0.43-0.75), and the discrimination to be satisfactory (Rat et al, 2006).
3. Western Ontario and McMaster Universities Arthritis Index (WOMAC): WOMAC is a disease-specific, self-administered health status measure that is widely used to assess the symptoms and physical disability for people with knee and/or hip OA. WOMAC has been translated into more than 65 different languages worldwide, in the current study it was translated by the researcher into the Arabic language, it has been validated for usage via telephone interviews, multimedia with audio-visual presentations, verbally spoken computer programs, and mobile phone applications. It is widely used in OA research especially to monitor the course of the disease or to determine the effectiveness of a variety of interventions (pharmacologic, surgical, physiotherapy etc.). It provides an excellent look at a patient's functional capacity and complements the more objective data provided by magnetic resonance imaging, arthroscopy, cartilage biopsy, and radiographs. It consists of 24 items divided into three subscales:

   * Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright
   * Stiffness (2 items): after first waking and later in the day
   * Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties.

   The Index is available in 5-point Likert (LK), 100mm visual analog (VA), and 11-point numerical rating (NR) scaling formats. On the Likert scale, each question had five alternatives where 0=no constraints or difficulties, 1 = slight, 2=moderate, 3=severe, 4= extreme. The highest score for each subscale on WOMAC on the Likert scale was 20 for pain, 8 for stiffness and 68 for physical function. The highest total score (96) denotes worse or more symptoms and the strongest physical constraints.
4. Knowledge, Attitude and Practice (KAP) questionnaire: to identify participants' knowledge about OA (what is KOA, symptoms, possible risk factors, complications, how to delay progression, management choices, and side effects), attitude towards non-surgical interventions and practices (nutritional habits, physical activity, treatment, and positions that worsen the condition or protect the knees).
5. Clinical assessment: the studied participants were subjected to clinical examination and anthropometric measurements (body mass index, waist and hip circumference).
6. Preintervention assessment of concentration of serum biomarker (IL-6) : A blood sample of 3cm was collected from all the participants after 12- hours fasting (to avoid the inflammatory effect of food) to measure inflammatory biomarkers (IL-6). This assessment was done on a sub sample of participants according to certain circumstances (as not receiving anti-inflammatory drugs in in the past 3 months and those who were adherent to the program of health education).

II) Health Education program Implementation: Nine educational sessions were held. In each session, 10-15 participants attended with total number of 109 participants. The session took 120 minutes.

1.The researcher provided successful aging topics using PowerPoint presentation mainly about 3 key messages:

1. What a regular physical activity and individualized exercise programs can reduce pain, prevent worsening and improve daily function in KOA.
2. The benefits of losing weight for overweight or obese patients, and the benefits of maintaining a healthy weight using diet changes and exercise.
3. Treatment of KOA and the fact that its symptoms can often be significantly reduced without the need of undergoing a surgery.

2.Rheumatologist and physiotherapist also provided messages about the following:

* What is KOA, its risk factors and symptoms, how it can vary greatly from person to person, and it is not an inevitable part of getting older
* Diagnostic methods and how joint damage on an X-ray does not indicate how much your osteoarthritis will affect you.
* Education about KOA treatment and medication intake (its side effects and how important to avoid the overuse of nonsteroidal anti-inflammatory drugs over the long term)
* How to protect your knees and the movements that should be avoided.
* A home-based exercise program which was created based on a literature review and consultation of experts aimed to increase lower-limb muscle strength, relieve pain, and balance. In addition, it was designed to strengthen the muscles supporting the knee, reduce knee stiffness, thus reducing stress on the knee joints. The program also worked on improving flexibility by stretching these muscles to improve range of motion and prevent injury. The exercises targeted the quadriceps, hamstrings, abductors, and adductors, as well as both the Gluteus Medius and Gluteus Maximus.

Before getting started with the exercises the participants were asked:

* Always warm up either with knee massage for 5 minutes or 5-10 minutes of low impact activity like walking in place or riding a stationary bicycle.
* Don't ignore the pain and feel free to ask the researcher if you have any pain while exercising.
* Ask questions if you are not sure how to do the exercise or how often to do it.
* Don't ignore stretching after strengthening exercises. The program consisted of three groups of exercises; each group lasted for two weeks. The participants performed the exercises twice daily according to their suitable time, but it was preferred early in the morning and before bedtime. Once the participant completed the exercises easily and without pain or cramps, he/she would go to the next new group of exercises.

The 1st group of exercises targeted and strengthened the muscles around the knee especially quadriceps muscle:

* Isometric quadriceps contraction
* Straight leg raises
* Lateral leg abduction
* Knee flexion in supine position
* Seated knee extension The participants started with 2 repetitions for each exercise, when the exercises got easier, they gradually increased the repetitions till they reached 10 repetitions twice daily.

The 2nd group of exercises worked on stretching the muscles of lower limbs

* Standing leg extension
* Standing hip abduction The main goal in this group of exercises was to gradually increase the time in which the muscle is under tension. The participants started with 5 seconds and 2 repetitions for each exercise till they reached 20-30 seconds with 5 repetitions by the end of the two weeks.

The 3rd group: The exercises worked on stretching and increasing the range of motion of front and back lower limb muscles (quadriceps muscle, hamstring muscle, gluteus muscle and calf muscles):

* Heel cord stretch
* Seated Leg raises
* Seated hip abduction
* Hamstring curls
* Seated leg extension The participants started with 5 seconds and 2 repetitions for each exercise till they reached 20-30 seconds with 5 repetitions by the end of the two weeks.

During the sessions, all the previous exercises were shown to the participants by a colleague and video recorded as well.

The researcher with the help of the supervisors designed an Educational Booklet after identifying the needs of the studied patients according to baseline health assessment. The booklet included information about osteoarthritis, risk factors, symptoms, diagnostic methods, how to delay its progression, healthy nutrition, importance of weight control and its influences, management of knee OA, physical activities, and home-based exercises with pictures of how to perform it. The booklet was distributed to the participants during the sessions.

3.WhatsApp groups were created for each group of exercises. Through each group, messages were distributed to summarize the content of the booklet. This is an easily accessible way to help them to follow the health education modifications and to keep them motivated to perform the home exercises every day, and to motivate each other. Exercises videos which were taped during the sessions were also sent in the group to remind them how to do each exercise correctly guided with the explanation in the booklet. This group also made it easier to the participants to contact the research team whenever they had any inquiry concerning exercises, lifestyle modifications.

4.Phone calls to follow up the participants and maximize their adherence to the health education program were done.

III) Post-intervention evaluation:

After six months of follow-up, this stage was carried out using WOMAC, OAKHQOL questionnaire, and KAP questionnaire to assess the effect of health education and lifestyle modification on the participants. Additionally, it was done to assess the activity, level of movement] and the degree of pain. Among the 104 participants who attended the health education sessions and finished the home exercise program, only 84 participants were able to fill the post-intervention questionnaires.

In the pre intervention, the mean scores of Il-6 for all participants were within normal (single and total), so there was no benefit of repeating it in the post intervention.

ELIGIBILITY:
Inclusion Criteria:

* KOA patients from both sexes.
* Age above 35 years old.
* One/both knee joint affection.

Exclusion Criteria:

* Other causes than OA for joint problems (e.g. hip fracture, chronic widespread pain, acute inflammatory joint disease, or cancer).
* Patients receiving physical therapy or intra-articular injection in the past 3 months.
* Total joint replacement or other surgery of the knee or hip within the past 3 months.
* Immunosuppressant intake in the past 3 months.
* Pregnancy, end stage disease or malignancy.

Ages: 36 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Assess the symptoms and physical disability, monitor the course of KOA, and determine the effectiveness of a variety of interventions | 6 months
  A Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a disease-specific, self-administered health status measure that is widely used. In the current study, WOMAC was translated by the researcher into the Arabic language. It consists of 24 items divided into three subscales: pain (5 items), stiffness (2 items), physical Function (17 items). The Index is available in 5-point Likert (LK), where 0=no constraints or difficulties, 1=slight, 2=moderate, 3=severe, 4= extreme. The highest score for each subscale on WOMAC on the Likert scale was 20 for pain, 8 for stiffness and 68 for physical function. The highest total score (96) denotes worse or more symptoms and the strongest physical constraints.
Measure QOL in KOA and assess the effect of health education and lifestyle modification | 6 months
  An Osteoarthritis Knee and Hip Quality of Life questionnaire (OAKHQOL) is a specific tool. In the current study, it was translated by the researcher into Arabic language. It has 43 items which fall into five domains: physical activity (16 items), mental health (13 items), pain (4 items), social support (4 items), social functioning (3 items), and three items are independent. Response to all items is by a Numerical Rating Scale (NRS) (0-10). A total score for each subscale is calculated by averaging the values for items of the same dimension and is normalized to a score from 0 (worst HRQOL) to 100 (best HRQOL).
Identify knowledge about KOA | 6 months
  Knowledge, Attitude and Practice (KAP) questionnaire to identify participants' knowledge about KOA: what is KOA, symptoms, possible risk factors, complications, how to delay progression, management choices, and side effects.
Identify attitude about KOA | 6 months
  Knowledge, Attitude and Practice (KAP) questionnaire to identify attitude towards non-surgical interventions.
Identify practices about KOA | 6 months
  Knowledge, Attitude and Practice (KAP) questionnaire to identify practices: (nutritional habits, physical activity, treatment, and positions that worsen the condition or protect the knees) and to assess the effect of health education and lifestyle modification on the participants.

SECONDARY OUTCOMES:
Sociodemographic data | 2 months
  Sociodemographic questionnaire: to gather information regarding participants age, gender, marital status, occupation, level of education, smoking habits, duration of the disease, medical history, and medications taken.
Clinical assessment | 2 months
  The studied participants were subjected to clinical examination and anthropometric measurements (body mass index, waist and hip circumference)
Measuring waist circumference | 2 months
  The studied participants were subjected to anthropometric measurements as waist circumference
Measuring hip circumference | 2 months
  The studied participants were subjected to anthropometric measurements as hip circumference
Serum IL-6 concentration assessment | 2 months
  This assessment was done on a sub sample of studied participants (n=76). A blood sample of 3cm was collected from all the participants after 12- hours fasting (to avoid the inflammatory effect of food) to measure inflammatory biomarkers (IL-6). This assessment was done on a sub sample of participants according to certain circumstances (as not receiving anti-inflammatory drugs in in the past 3 months and those who were adherent to the program of health education).
Measuring body mass index | 2 months
  The studied participants were subjected to anthropometric measurements as body mass index by measuring Weight and Height

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Centre, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No